CLINICAL TRIAL: NCT00000435
Title: A Clinical Trial of Shared Epitope Peptides in Rheumatoid Arthritis (RA)
Brief Title: dnaJ Peptide for Relieving Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01 AR92241; NIAMS-042
Record Dates: First submitted 2000-01-21; First posted 2000-01-24 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-07

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Immune Modulation; Oral Tolerance; Peptide; dnaJ
MeSH Terms: conditions — Arthritis, Rheumatoid

ARMS (2):
- A (Placebo Comparator): Subjects randomized to arm A received 25mg/day po of placebo
  Interventions: Drug: None-placebo
- B (Active Comparator): Subjects randomized to Arm B received 25mg/day po of peptide dnaJP1
  Interventions: Drug: dnaJ peptide

INTERVENTIONS:
Drug: dnaJ peptide — dnaJP1 was taken in pill form at 25mg/day for 6 months
  Arms: B
Drug: None-placebo — placebo was taken in pill form at 25mg/day for 6 months
  Arms: A

SUMMARY:
A small protein called dnaJ peptide may help people with rheumatoid arthritis (RA) by preventing their immune system cells from attacking their own tissues. The purpose of this study is to determine if small amounts of dnaJ peptide can "re-educate" immune cells in people with RA so that the cells stop attacking joint tissues.

DETAILED DESCRIPTION:
Immune modulation is a promising new approach for the treatment of RA. Studies have shown that immune cells in the joints of people in the early stages of RA react strongly against dnaJ peptides from bacteria. These immune cells may also cross-react with human dnaJ peptides in the joints to cause inflammation. dnaJ may help RA by "re-educating" the immune system and dampening the abnormal inflammatory immune response in RA.

This study will last 7 months. Participants will be randomly assigned to receive either dnaJ or placebo by mouth. At screening, participants will have medical history, physical, and medication assessment. At screening, at 6 study visits every month after the start of treatment, and at 1 month follow-up, participants will have a joint exam, blood and urine collection, and will fill out a questionnaire about their condition.

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis as defined by the revised American College of Rheumatology (ACR) 1987 criteria. Evidence of active disease will be based on at least six swollen or nine tender joints.
* Diagnosis of rheumatoid arthritis of less than 5 years
* Reactivity to dnaJ
* Agree to use acceptable methods of contraception
* Able to understand and sign informed consent

Exclusion Criteria:

* Patients taking more 7.5 mg of prednisone or disease modifying agents other than hydrochloroquine or sulfasalazine (i.e., gold, penicillamine, azathioprine, cyclophosphamide, methotrexate, cyclosporine, or anti-TNF agents)
* Serum creatinine greater than 1.5 mg/dl
* SGOT less than SGPT
* Alkaline phosphatase greater than 2 times age/sex adjusted normal values
* Hematocrit of less than 30
* Platelets less than 130,000
* History of lymphoma
* Any active malignancy or cancer requiring treatment in the last 5 years, except for nonmelanoma skin cancers and carcinoma of the cervix in situ
* Medical or psychiatric condition or active serious infection
* Pregnant or breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 1999-09; Study Completion 2004-09

PRIMARY OUTCOMES:
Area under the curve or 'AUC' obtained by adding 0 for no response and 1 for an ACR 20 response for visits on Day 112, 140, and 168 | time points 112, 140 and 168 of the 6-month trial

SECONDARY OUTCOMES:
Day 112 ACR 20 score | Visit day 112 of the 6-month trial

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Albani, MD, Principal Investigator — University of California, San Diego
Locations (8):
- United States (8):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - University of California, Irvine Medical Center, Orange, California
  - Stanford University, Palo Alto, California
  - Denver Arthritis Center, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Guthrie Clinic, Sayre, Pennsylvania
  - Virginia Mason Research Center, Seattle, Washington

REFERENCES:
- [Background] Prakken BJ, Samodal R, Le TD, Giannoni F, Yung GP, Scavulli J, Amox D, Roord S, de Kleer I, Bonnin D, Lanza P, Berry C, Massa M, Billetta R, Albani S. Epitope-specific immunotherapy induces immune deviation of proinflammatory T cells in rheumatoid arthritis. Proc Natl Acad Sci U S A. 2004 Mar 23;101(12):4228-33. doi: 10.1073/pnas.0400061101. Epub 2004 Mar 15. PMID 15024101
- [Derived] Koffeman EC, Genovese M, Amox D, Keogh E, Santana E, Matteson EL, Kavanaugh A, Molitor JA, Schiff MH, Posever JO, Bathon JM, Kivitz AJ, Samodal R, Belardi F, Dennehey C, van den Broek T, van Wijk F, Zhang X, Zieseniss P, Le T, Prakken BA, Cutter GC, Albani S. Epitope-specific immunotherapy of rheumatoid arthritis: clinical responsiveness occurs with immune deviation and relies on the expression of a cluster of molecules associated with T cell tolerance in a double-blind, placebo-controlled, pilot phase II trial. Arthritis Rheum. 2009 Nov;60(11):3207-16. doi: 10.1002/art.24916. PMID 19877047